CLINICAL TRIAL: NCT07153120
Title: Evaluation of Erich Arch Bars, IMF Screws and Hybrid Arch Bars in the Management of Mandibular Fractures: A Randomized Clinical Study
Brief Title: Erich Arch Bars, IMF Screws and Hybrid Arch Bars in the Management of Mandibular Fractures
Acronym: Jaw Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Zead Ahmad Khaled Murad Alkurdi, Clinical demonstrator at oral and maxillofacial surgery department, faculty of dentistry, Mansoura University, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS.25.04.16
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-04

CONDITIONS: Mandibular Fractures
Keywords: Arch bars; Erich arch bars; Hybrid arch bars; Mandibular fractures; IMF Screws; MMF; IMF; Maxillomandibular Fixation; Jaw fractures; Maxillofacial Trauma; Mandibulomaxillary Fixation
MeSH Terms: conditions — Mandibular Fractures; Jaw Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HAB Group (Experimental)
  Interventions: Device: Hybrid Arch Bars
- EAB Group (Experimental)
  Interventions: Device: Erich Arch Bars
- IMF Screws Group (Experimental)
  Interventions: Device: IMF Screws

INTERVENTIONS:
Device: Erich Arch Bars — Stainless steel plates with hooks for wire placement are adapted over the facial aspect of teeth so the wires would be inserted to go around the necks of teeth (circumdental wiring), then both maxillary and mandibular plates are ligated to each other in order to achieve MMF.
  Arms: EAB Group
Device: Hybrid Arch Bars — Screw retained titanium plates with hooks for wires are adapted properly then self drilling self locking screws will be drilled in between roots of teeth to avoid injury, after fixation both jaws will be wired to accomplish MMF
  Arms: HAB Group
Device: IMF Screws — A total of four self drilling screws two in the maxilla and the other two in the mandible will be inserted in the bone above and below teeth roots apices to avoid injury, to be ligated to each other in a vertical and an X pattern to achieve MMF.
  Arms: IMF Screws Group

SUMMARY:
Treatment options of mandibular fractures can be accomplished with either closed treatment or open reduction internal fixation (ORIF). Maxillomandibular fixation (MMF) refers to any method used to secure the maxilla and mandible in proper dental occlusion. MMF is a standard component of mandibular fracture management essential for closed treatment and commonly used du ring ORIF. Its three main principles are to establish occlusion, provide stability, and immobilize the jaws.

DETAILED DESCRIPTION:
An abundance of modalities used for establishing MMF have been reported in the literature. Traditionally, Ivy eyelets wiring, Risdon wiring, metal splints, acrylic splints and Erich arch bars are used. Progressively, new techniques such as Intermaxillary Fixation (IMF) screws, wiring around single tooth with tight contacts, use of 2 miniplates, use of zip ties, use of bondable buttons and 2 looped wires have been developed to expedite securement of MMF.

The conventional MMF procedure uses arch bars of malleable strips of steel-bearing hooks, also known as Erich arch bars (EABs), allowing hands-free achievement and maintenance of excellent intraoperative occlusion with reproducibility.

However, the placement of Erich arch bars (EABs) fixated to the dentition with circumdental stainless-steel wires has been the standard practice for MMF for or during the repair of mandibular fractures for many decades.

Most of these techniques are limited in the setting of poor dentition or in patients who are partially edentulous, in addition of being time consuming, and are associated with risks of mucosal, dental, and needlestick injuries.

A hybrid arch bar (HAB) for MMF has been introduced to overcome some disadvantages of conventional arch bars. The HAB differs from the EAB because they are secured directly to the alveolar bone with screws rather than using teeth for anchorage.

Some authors suggest that IMF screws are less time consuming, provide better oral hygiene and reduce the risk of needle stick injury. Conversely, IMF screws have been associated with teeth root damage and screw loosening which can compromise MMF. Despite these disadvantages, IMF screws remain a recommended alternative to traditional arch bars for management of maxillofacial trauma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mandibular fracture indicated for MMF. (Favorable fractures, minimally displaced).
2. Patients with an age range from 18:50 years old.
3. Patients free from any systemic diseases.

Exclusion Criteria:

1. Patients that are not willing to participate in this clinical trial.
2. Edentulous patients or those with inadequate dentition for occlusal guidance
3. Pathological fractures.
4. Patients with absolute or relative contraindications to MMF (e.g. pregnancy, mental disorders and systemic diseases).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Occlusal Stability (evaluated clinically) | Four to six weeks
Time taken to apply fixation device | Four to six weeks

SECONDARY OUTCOMES:
Wire retightening frequency | Four to six weeks
Soft tissue evaluation (oral hygiene scores using Gingival Index) | Four to six weeks
Patient acceptance and hardware tolerability (evaluated using Visual Analog Scale (VAS) | Four to six weeks
Fracture union (evaluated radiographically using CBCT and Panoramic radiographs). | Four to six weeks
Complications (e.g., iatrogenic injuries, displacement, splaying) | Four to six weeks
Gloves perforation incidence | Four to six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided